CLINICAL TRIAL: NCT02632903
Title: Intravenous Zoledronic Acid for the Treatment of Osteoporosis and Osteonecrosis in Children With Leukemia: A Pilot Study
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: While the clinical need for and the scientific merit remain valid, this regulated drug trial was not feasible logistically due to limited funds.
Sponsor: Children's Hospital of Eastern Ontario (Other)
Responsible Party: Principal Investigator, Dr. Leanne Ward, MD, Children's Hospital of Eastern Ontario
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZA8DEC2015
Record Dates: First submitted 2015-12-15; First posted 2015-12-17 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Osteoporosis; Osteonecrosis; Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Osteoporosis; Osteonecrosis; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intravenous Zoledronic Acid (Experimental): Intravenous Zoledronic Acid 0.025mg/kg at baseline and 6 months
  Interventions: Drug: Zoledronic acid

INTERVENTIONS:
Drug: Zoledronic acid

SUMMARY:
This study explores the effect of zoledronic acid on incident vertebral fractures and osteonecrotic lesions in children recently diagnosed with acute lymphoblastic leukemia.

ELIGIBILITY:
Inclusion Criteria:

1. Subject or subject's legally acceptable representative has provided informed consent.
2. Children aged 8 to 16 years at the time of enrolment with a confirmed diagnosis of acute lymphoblastic leukemia (ALL).
3. Children with vertebral fractures or osteonecrotic lesions according to the following criteria:

   1. children with vertebral fractures on lateral spine x-ray and/or osteonecrotic lesions on MRI of the hips and/or knees identified through routine clinical screening at least 8 weeks following chemotherapy initiation OR
   2. children with vertebral fractures on lateral spine x-ray and/or osteonecrotic lesions of the hips and/or knees on MRI that are identified at any time in the first 12 months after chemotherapy initiation following presentation with back pain (in the case of vertebral fractures, identified by lateral spine x-rays) and/or hip pain (in the case of osteonecrotic lesions, identified by MRI) and/or knee pain (in the case of osteonecrotic lesions, identified by MRI).

Exclusion Criteria:

1. Any child for whom the treating physician feels participation is not advised.
2. Prior treatment with an osteoporosis agent (e.g. bisphosphonate).
3. Co-morbidities affecting musculoskeletal health (e.g. cerebral palsy).
4. Children with renal failure (eGFR<60ml/min/1.73m2).
5. Children with untreated vitamin D deficiency (vitamin D <50nmol/L).
6. Children with hypocalcemia.
7. Children planning dental procedures and/or dental surgery during the course of the study.
8. Children with asthma who are acetylsalicylic acid (ASA) sensitive.
9. Children with a documented history of atrial fibrillation.
10. Currently pregnant or planning a pregnancy during the study.
11. Currently breastfeeding or planning on breastfeeding during the study.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-10; Primary Completion 2018-03 (Estimated); Study Completion 2018-08-20 (Actual)

PRIMARY OUTCOMES:
To assess the effect of zoledronic acid on preventing incident vertebral fractures | 15 months post-diagnosis (12 months after baseline visit)
  To assess the effect of zoledronic acid on preventing incident vertebral fractures as measured by lateral spine radiographs at 15 months post-diagnosis compared to baseline (with baseline occurring 3 months post-diagnosis). An incident vertebral fracture on lateral spine radiographs will be defined as a new fracture (Genant Grade 1 or more) in a previously normal vertebral body, or worsening of an existing fracture (increase in Genant Grade by at least 1) on the follow-up x-ray that takes place 12 months after the first dose.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes